CLINICAL TRIAL: NCT02450461
Title: Exhaled Breath Analysis by Secondary Electrospray Ionization (SESI-MS) in Patients With Asthma
Brief Title: Breath Analysis in Asthma
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2015-0148
Record Dates: First submitted 2015-04-29; First posted 2015-05-21 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Asthma; Exhaled Breath; Mass Spectrometry
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asthma: 20 patients with asthma
  Interventions: Other: no intervention
- Controls: 20 control subjects with no apparent lung disease and normal lung function testing. Matched for gender, age and smoking history.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The purpose of this study is to answer the question whether a disease-specific profile of breath in patients with asthma can be detected by an untargeted metabolomic study using exhaled breath analysis by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed asthma. Diagnosis of asthma is made with episodic chest symptoms and a documented reversibility of at least 12% and/or 200 ml in FEV1 after 200 ug of inhaled salbutamol or airway hyperresponsiveness in the case of normal lung function testing (PC20 methacholine < 4mg/ml) at the time of diagnosis.
2. Age between 18 and 80 years at study entry.
3. Healthy controls: never-smokers, normal spirometry (baseline FEV1 > 85% predicted and FEV1/FVC greater than 0.7).

Exclusion Criteria:

1. Asthma exacerbation within the last 6 weeks, defined as worsening of asthma symptoms requiring a change in therapy by a physician or a change in regular asthma therapy (including short course of oral corticosteroids)
2. Any lung disease other than asthma.
3. Acute inflammatory disease (e.g. common cold) within the last 4 weeks.
4. Regular intake of oral steroids.
5. Active smoking habits / positive history of smoking.
6. Acute or chronic hepatic disease.
7. Renal failure or renal replacement therapy.
8. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from asthma will be included according to the predefined inclusion and exclusion criteria.
  Healthy controls will be recruited from the general population by printed flyers, newspaper advertisements and personal communication.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the asthma specific mass spectrometric profile of VOCs of exhaled breath analysis (markers of asthma in exhaled breath) | 1 day, single measurement, no follow up

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Switzerland